CLINICAL TRIAL: NCT00056641
Title: An Open Label, Randomized, Parallel-group Pharmacokinetics Trial of Tipranavir / Ritonavir (TPV/RTV), Alone or in Combination With RTV-boosted Saquinavir (SQV), Amprenavir (APV), or Lopinavir (LPV), Plus an Optimized Background Regimen, in Multiple Antiretroviral (ARV) Experienced Patients.
Brief Title: Dual Boosted - Protease Inhibitor (PI) Pharmacokinetics (PK) Trial (Tipranavir / Ritonavir) in Highly Treatment-experienced HIV-1 Infected Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1182.51
Record Dates: First submitted 2003-03-19; First posted 2003-03-21 (Estimated); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — tipranavir; Ritonavir; Saquinavir; amprenavir; Lopinavir

INTERVENTIONS:
Drug: tipranavir
Drug: ritonavir
Drug: saquinavir
Drug: amprenavir
Drug: lopinavir

SUMMARY:
This is an open-label, randomized, parallel group pharmacokinetics trial of tipranavir/ritonavir (TPV/RTV), alone or in combination with RTV-boosted saquinavir (SQV), amprenavir (APV) or lopinavir (LPV), plus an optimized background regimen, in multiple antiretroviral (ARV) experienced HIV-1 patients.

The primary objective is to determine the safety and pharmacokinetics of:

TPV/RTV given with an optimized background regimen (OBR) and TPV/RTV given in combination with saquinavir, amprenavir, or Kaletra® and an optimized background regimen (OBR).

ELIGIBILITY:
Inclusion criteria:

* Signed informed consent prior to trial participation.
* Human Immunodeficiency Virus type 1 (HIV-1) infected males or females ≥18 years of age.
* Acceptable laboratory screening values in Trial 1182.12 (RESIST 1) or 1182.48 (RESIST 2), excluding genotype.
* Genotypic resistance report from screening visit of study RESIST 1 or RESIST 2 indicating at least three mutations at protease codons 33, 82, 84, and 90.
* At least 3 consecutive months experience taking ARVs from each of the classes of Nucleoside reverse transcriptase inhibitors (NRTI), Non-nucleoside reverse transcriptase inhibitor 1 (NNRTI), and Protease Inhibitor (PI) at some point in treatment history, with at least 2 PI-based regimens, one of which must be part of the current regimen, and current PI-based Anti-retroviral (ARV) medication regimen for at least 3 months prior to randomization.
* HIV-1 viral load ≥1000 copies/mL at screening.
* Further inclusion criteria apply.

Exclusion criteria:

* Anti-retroviral (ARV) medication naïve.
* Patients on recent drug holiday, defined as off ARV medications for at least 7 consecutive days within the last 3 months.
* Female patients of child-bearing potential who:

  * have a positive serum pregnancy test at screening or during the study,
  * are breast feeding,
  * are planning to become pregnant,
  * are not willing to a use barrier method of contraception, or
  * require ethinyl estradiol administration.
* Prior tipranavir use.
* Use of investigational medications within 30 days before study entry or during the trial.
* Further exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328
Dates: Start 2003-02-18 (Actual); Primary Completion 2004-01-27 (Actual)

PRIMARY OUTCOMES:
Change of the 2nd Protease Inhibitor (PI) (APV, LPV. SQV) mean concentration (C12h) | Day 14 to Day 28
Occurrence of adverse events; Proportion of patients with laboratory abnormalities; Proportion of patients with SAEs | week 4

SECONDARY OUTCOMES:
Mean concentration (C12h) of TPV (TPV/r group); Mean concentration (C12h) of RTV (TPV/r group) | Week 1 and 2
Mean concentration (C12h) of TPV (PI/TPV/r group); Mean concentration (C12h) of RTV (PI/TPV/r group) | Week 3 and 4
Assessment of patient adherence | Week 1 to 4
Area under the Curve (AUC(0-12h)) of the 2nd PI (APV, LPV. SQV); Maximum concentration (Cmax) of the 2nd PI (APV, LPV. SQV); Concentration (C12h) of the 2nd PI (APV, LPV. SQV) | week 2 and 4
Change in AUC(0-12h) of TPV from week 2; Change in Cmax of TPV from week 2; Change in C12h of TPV from week 2 | week 4
Change in AUC(0-12h) of RTV from week 2; Change in Cmax of RTV from week 2; Change in C12h of RTV from week 2 | week 4
AUC(0-12h) of RTV; Cmax of RTV; C12h of RTV | week 2 and 4
Change in viral load; Proportion of virologic responders | week 2, 4, 8, 16 and 24

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim Study Coordinator, Study Chair — Boehringer Ingelheim
Locations (109):
- United States (34):
  - Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - Boehringer Ingelheim Investigational Site, Berkeley, California
  - Boehringer Ingelheim Investigational Site, Fountain Valley, California
  - Boehringer Ingelheim Investigational Site, Los Angeles, California
  - Boehringer Ingelheim Investigational Site, San Francisco, California
  - Kaiser Permanente Medical Center, San Francisco, California
  - San Francisco VAMC, San Francisco, California
  - Boehringer Ingelheim Investigational Site, Norwalk, Connecticut
  - Washington DC VA Medical Center, Washington D.C., District of Columbia
  - North Broward Hospital District, Fort Lauderdale, Florida
  - Boehringer Ingelheim Investigational Site, Fort Myers, Florida
  - Boehringer Ingelheim Investigational Site, Miami, Florida
  - Boehringer Ingelheim Investigational Site, Orlando, Florida
  - Boehringer Ingelheim Investigational Site, Sarasota, Florida
  - Boehringer Ingelheim Investigational Site, Tampa, Florida
  - Boehringer Ingelheim Investigational Site, Vero Beach, Florida
  - Boehringer Ingelheim Investigational Site, Atlanta, Georgia
  - Mercer University School of Medicine, Macon, Georgia
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Boehringer Ingelheim Investigational Site, Boston, Massachusetts
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Boehringer Ingelheim Investigational Site, Springfield, Massachusetts
  - Henry Ford Hospital, Detroit, Michigan
  - Boehringer Ingelheim Investigational Site, Santa Fe, New Mexico
  - Albany Medical College, Albany, New York
  - Boehringer Ingelheim Investigational Site, New York, New York
  - University of New York, Stony Brook, Stony Brook, New York
  - Duke University Medical Center, Durham, North Carolina
  - Boehringer Ingelheim Investigational Site, Huntersville, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - UT Southwestern, Dallas, Texas
  - Boehringer Ingelheim Investigational Site, Houston, Texas
  - Boehringer Ingelheim Investigational Site, Annandale, Virginia
  - Boehringer Ingelheim Investigational Site, Tacoma, Washington
- Australia (2):
  - Boehringer Ingelheim Investigational Site, Darlinghurst, New South Wales
  - St. Vincent's Hospital, Darlinghurst, New South Wales
- Belgium (3):
  - Instituut Tropische Geneeskunde, Antwerp
  - Centre Hospitalier Universitaire St. Pierre, Brussels
  - U.Z. Gent, Ghent
- Canada (7):
  - McMaster University Medical Centre, Hamilton, Ontario
  - Boehringer Ingelheim Investigational Site, Toronto, Ontario
  - Canadian Immunodeficiency Research Collaborative Inc., Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - McGill University Health Centre, Suite A5-140, Monteal, Quebec
  - Boehringer Ingelheim Investigational Site, Montreal, Quebec
  - Montreal Chest Institute - McGill University Health Centre, Montreal, Quebec
- Denmark (3):
  - Hvidovre Hospital, Hvidovre
  - Rigshospitalet, København Ø
  - Odense Universitetshospital, Odense C
- France (14):
  - Hôpital Pellegrin, Bordeaux
  - Hôpital Côte de Nacre, Caen
  - Hôpital Antoine Beclère, Clamart
  - Hôpital de l'Hôtel Dieu, Lyon
  - Hôpital Hôtel Dieu, Nantes
  - Hôpital de l'Archet, Nice
  - Hôpital Bichat Claude Bernard, Paris
  - Hôpital de la Pité Salpêtrière, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Saint Antoine, Paris
  - Hôpital de Pontchaillou, Rennes
  - Hôpital civil, Strasbourg
  - Hôpital brabois, Vandœuvre-lès-Nancy
  - Hôpital Paul Brousse, Villejuif
- Germany (21):
  - Boehringer Ingelheim Investigational Site, Aachen
  - Epimed GmbH, Berlin
  - Universitätsklinikum Charité, Berlin
  - Medizinische Universitätsklinik Bonn, Bonn
  - Klinik I für Innere Medizin der, Cologne
  - Boehringer Ingelheim Investigational Site, Düsseldorf
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Universitätsklinik Erlangen-Nürnberg, Erlangen
  - Universitätsklinikum Essen, Essen
  - Klinikum der Johann Wolfgang Goethe-Universität, Frankfurt am Main
  - Boehringer Ingelheim Investigational Site, Freiburg im Breisgau
  - Universitätsklinkum Freiburg, Freiburg im Breisgau
  - ifi Institut für interdisziplinäre Infektiologie, Hamburg
  - Universitätsklinik Hamburg-Eppendorf, Hamburg
  - Med. Hochschule Hannover, Hanover
  - Universitätsklinikum Heidelberg, Heidelberg
  - Facharzt für Innere Medizin,, Mannheim
  - Boehringer Ingelheim Investigational Site, München
  - Medizinische Poliklinik, München
  - Klinium Natruper Holz, Osnabrück
  - Boehringer Ingelheim Investigational Site, Stuttgart
- Greece (9):
  - 1st Social Insurance Foundation (IKA) Pentelis, Athens
  - Andreas Syggros Hosp., Athens
  - Evangelismos Hospital, Athens
  - General Hospital "G. Gennimatas", Athens
  - Korgialenio-Benakio-Hellenic Red Cross General Hospital, Athens
  - Sismanoglio Hospital, Athens
  - University Hospital of Patras, Pátrai
  - "Tzanio" Hospital, Piraeus
  - AHEPA Hospital, Thessaloniki
- Italy (2):
  - Fondazione S. Raffaele del Monte Tabor, Milan
  - Ospedale Amedeo di Savoia, Torino
- Netherlands (4):
  - OLVG, Amsterdam
  - Slotervaart Hospital, Amsterdam
  - Erasmus Medical Centre, Rotterdam
  - Medical Centre Haaglanden, The Hague
- Portugal (4):
  - Hospital Condes Castro Guimarães, Cascais
  - Hospitais da Universidade de Coimbra, Coimbra
  - Department of Infeccious Diseases, Lisbon
  - Hospital de São João, Porto
- Switzerland (3):
  - Universitätsspital Basel, Basel
  - Kantonsspital St. Gallen, Sankt Gallen
  - Universitätsspital Zürich, Zurich
- United Kingdom (3):
  - Royal Free Hospital, London
  - SSAT/Crusaid Institute, London
  - St Mary's Hospital, London